CLINICAL TRIAL: NCT01552967
Title: A Phase II Trial Evaluating a Modified Regimen of Oxaliplatin and Capecitabine in First-Line Treatment of Metastatic Colorectal Adenocarcinoma
Brief Title: Efficacy and Safety Study of a Modified XELOX Regimen in First-Line Treatment of Metastatic Colorectal Adenocarcinoma
Acronym: mXELOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHMO-01
Record Dates: First submitted 2012-03-05; First posted 2012-03-13 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Adenocarcinoma
Keywords: Colorectal cancer; Adenocarcinoma; XELOX
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine — Oxaliplatin 85mg/m2 D1 and capecitabine 1g/m2 BID D1-D10, repeat every two weeks.
  Efficacy will be evaluated every three cycles.

SUMMARY:
This is an open-label, phase II study to evaluate the efficacy and safety of a modified regimen of oxaliplatin and capecitabine on metastatic colorectal adenocarcinoma in the first-line therapy.

DETAILED DESCRIPTION:
Primary endpoint: Overall Response Rate

Secondary endpoint: Time to progression, overall survival, safety data

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Patients with histologically or cytologically confirmed stage IV colorectal adenocarcinoma whose ECOG performance status are 0-2;
* Presence of measurable disease by radiographic study (including CT or MRI scan, or chest x-ray) or physical examination;
* At least 3 weeks since last major surgery;
* At least 12 months since last adjuvant chemotherapy;
* At least 6 weeks since prior radiotherapy providing that the extent and site of radiotherapy fields are such that marked bone marrow suppression is NOT expected;
* Patients who have received palliative radiotherapy must have recovered from any reversible toxic effects e.g. nausea and vomiting caused by radiation of fields;
* Patients with reproductive potential must use effective BC;
* Required Screening Laboratory Criteria:

  * Hemoglobin 90g/L
  * WBC 3.5 x 109/L
  * Neutrophils 1.5 x 109/L
  * Platelets 100 x 109/L
  * Creatinine 133 umol/L and creatinine clearance 60 mL/min
* A probable life expectancy of at least 6 months;

Exclusion Criteria:

* Brain metastases;
* Female of childbearing potential, pregnancy test is positive;
* Concomitant malignancies or previous malignancies other than colorectal cancer within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or low grade prostate cancer;
* Active infection;
* Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to extreme risk;
* Sexually active patients refusing to practice adequate contraception;
* Patients with conditions which might affect absorption of an oral drug (for example intermittent obstruction) unless discussed and agreed with principal investigator;
* History of grade 3 or 4 toxicity to fluoropyrimidines;
* Pre-existing neuropathy ≥ NCI CTC grade 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate according to RECIST 1.1 | One year

SECONDARY OUTCOMES:
Time to progression | One year
overall survival | One Year
Safety data of this regimen | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiao, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China